CLINICAL TRIAL: NCT02041052
Title: Phase Two Randomized Study of The Size of the Gastric Remnant as Determinant for Delayed Gastric Emptying After Whipple Resection.
Brief Title: The Size of the Gastric Remnant as Determinant for Delayed Gastric Emptying After Whipple Resection.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to insufficient inclusion rate.
Sponsor: Karolinska University Hospital (Other)
Collaborators: Ralf Segersvärd (Unknown); Afshin Noorani (Unknown); John Blomberg (Unknown)
Responsible Party: Principal Investigator, Lars Lundell, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/1262-31/3; 2011/1262-31/3 (Other: Swedish Ethic Committee)
Record Dates: First submitted 2013-12-10; First posted 2014-01-20 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: 50 % Reduction of Delayed Gastric Emptying

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Whipple procedure (Active Comparator): Conventional Whipple procedure
  Interventions: Procedure: Conventional whipple procedure
- Subtotal gastrectomy added to whipple procedure. (Experimental): Subtotal gastrectomy added to Whipple procedure.
  Interventions: Procedure: Subtotal gastrectomy as an adjunct to traditional whipple procedure.

INTERVENTIONS:
Procedure: Subtotal gastrectomy as an adjunct to traditional whipple procedure. — Subtotal gastrectomy as an adjunct to traditional whipple procedure.
  Arms: Subtotal gastrectomy added to whipple procedure.
Procedure: Conventional whipple procedure — All patients undergoing whipple procedure without risk for pancreaticojejunal anastomosis leakage.
  Arms: Conventional Whipple procedure

SUMMARY:
A small gastric remnant after whipple resection improves gastric emptying and therefore prevents the development of delayed gastric emptying.

DETAILED DESCRIPTION:
Every patient submitted to a whipple resection and at the same time present with characteristics suggestive of minimal risk for leakage from the pancreaticojejunostomy will be included in the study. At the time of reconstruction the patient will be randomized to either conventional size of the stomach or to a subtotal gastrectomy containing a small upper gastric pouch only.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing whipple procedure with preoperative assignment as low risk for leakage from the pancreaticojejunal anastomosis.

* Signed informed consent.

Exclusion Criteria:

* High and intermediate risk pancreaticojejunal anastomosis. Unwillingness to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Postoperative delayed gastric emptying | Postoperative recovery period in days (on an average <20 days)
  During the postoperative phase the patient will be followed daily with assessment of symptoms suggestive of delayed gastric emptying.

SECONDARY OUTCOMES:
Quality of life | during three first postoperative months
  Quality of life measured by use of scientifically validated instruments.
Postoperative hospital stay | In hospital stay in days (on an average <20 days)
  Time in days from the operation to discharge from hospital.
Total Gastric emptying as measured by the paracetamol test | three months postoperatively
  Paracetamol orally ingested together with chocolate biscuits whereafter peripheral venous blood concentrations of paracetamol are determined. Blood samples taken at baseline and every 15 minutes after paracetamol ingestion during the first hour and then every 30 minutes for an hour.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lundell, professor, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital Gastrocentrum, Stockholm, Sweden